CLINICAL TRIAL: NCT04375943
Title: Clinical and Echocardiographic Management of Patients With Chronic Heart Failure and Type 2 Diabetes Mellitus: the SCODIAC Follow up Study
Brief Title: Clinical and Echocardiographic Management of Patients With Heart Failure and Diabetes: SCODIAC Follow up Study
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Oliviero Ugo, Principal investigator, Federico II University
Other Study IDs: FedericoIIArcaAmd
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Diabetes; Heart Failure
Keywords: diabetes; heart failure; ejection fraction
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure | interventions — Hypoglycemic Agents; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic HF-pEF patients: It is composed of 136 HF diabetic patients with preserved Ejection Fraction (HF-pEF) (>45%).
  Interventions: Drug: Antidiabetic
- diabetic HF-rEF patients: It is composed of 270 HF diabetic patients with reduced EF (HF-rEF) (≤45%).
  Interventions: Drug: Antidiabetic

INTERVENTIONS:
Drug: Antidiabetic — Verify whether the use of innovative antidiabetic therapies could modify echocardiographic parameters and influence cardiological therapy
  Other Names: SGLT2 inhibitors, gliflozins, echocardiography.

SUMMARY:
The study has been carried out to determine diagnostic and therapeutic pathways in a group of HF diabetic patients and to verify whether the use of innovative antidiabetic therapies could modify echocardiographic parameters and influence cardiological therapy.

DETAILED DESCRIPTION:
406 patients affected with heart failure and Type 2 Diabetes Mellitus, referred to Cardiologists and Diabetologists of pertaining healthcare districts in Campania, and followed for at least one year between 2018 and 2019, were enrolled in this retrospective study and divided in Group A, composed of 136 HF diabetic patients with preserved Ejection Fraction (HF-pEF) (>45%) and Group B, formed of 270 HF diabetic patients with reduced EF (HF-rEF) (≤45%). All patients had performed periodic clinical evaluations and an echocardiographic exam every 12 months. Anthropometric parameters, HF etiology, co-morbidities, complications and ongoing therapies were collected.

ELIGIBILITY:
Inclusion Criteria:

* age at least 65 years
* presence of chronic HF, defined as a stable clinical syndrome with typical symptoms and signs and echocardiographic evidence of cardiac involvement
* New York Heart Association (NYHA) class II-III
* diagnosis of T2DM from at least 2 years

Exclusion Criteria:

* cardiac surgery performed during the last year
* age less than 65 years
* significant valvulopathies
* malignant neoplasms
* advanced chronic kidney disease

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A total of 406 patient with HF and T2DM, referred to ARCA Cardiologists from 17 healthcare districts in Campania and to AMD Physicians from 8 Antidiabetic Centers and followed for at least one year between 2018 and 2019, were enrolled.
Sampling Method: Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol, LDL, HDL Triglycerides, Creatinine | 12 months
  mg/dl
B-type natriuretic peptide (BNP) | 12 months
  pmol/m
HbA1c | 12 months
  mmol/L
Ejection Fraction | 12 months
Left Ventricular End-Diastolic Volume Index (LV-EDVi), Left Ventricular End-Systolic Volume Index (LV-ESVi), Left Atrial Volume Index (LAVi) | 12 months
  ml/m2
E velocity, A velocity,E' velocity | 12 months
  m/sec

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Oliviero, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided